CLINICAL TRIAL: NCT00726908
Title: Intramuscular Lipid and Insulin Action:Ethnic Aspects
Acronym: QuEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara Gower, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: F070322005; R01DK067538 (NIH)
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: Obesity; diet; carbohydrate; insulin
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Low carbohydrate — 43% CHO

SUMMARY:
High levels of the hormone insulin are associated with risk for heart disease and diabetes, and may make it hard to lose weight. The types of food eaten may affect insulin levels. The purpose of this study is to determine if manipulation of dietary carbohydrate content improves insulin sensitivity (Si), augments weight loss, and promotes weight loss maintenance in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

Overweight, age 21-50 years,Women must be premenopausal, Normal glucose tolerance, weight stable for at least 6 months with a weight change no greater than 5 lbs.

Exclusion Criteria:

Exclusion criteria were type 1 or type 2 diabetes, polycystic ovarian disease, BMI <26.5 or weight >300 pounds, weight change >5 pounds in last 6 months, regular exercise >2 hours per week, pregnancy, currently breastfeeding, cholesterol medications, any disorders of glucose or lipid metabolism, use of medication that could affect body composition or glucose metabolism (including oral contraceptives and blood pressure medications), current use of tobacco, use of illegal drugs in last 6 months, history of hypoglycemic episodes, major food allergies or food dislikes, women with inconsistent or absence of monthly menstrual cycles, and a medical history that counter-indicated inclusion in the study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | IVGTT and minimal model

SECONDARY OUTCOMES:
Weight loss | Weight loss over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Gower, PhD, Principal Investigator — Univ. Alabama Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Morrison SA, Goss AM, Azziz R, Raju DA, Gower BA. Peri-muscular adipose tissue may play a unique role in determining insulin sensitivity/resistance in women with polycystic ovary syndrome. Hum Reprod. 2017 Jan;32(1):185-192. doi: 10.1093/humrep/dew279. Epub 2016 Nov 8. PMID 27827322
- [Derived] Gower BA, Goss AM. A lower-carbohydrate, higher-fat diet reduces abdominal and intermuscular fat and increases insulin sensitivity in adults at risk of type 2 diabetes. J Nutr. 2015 Jan;145(1):177S-83S. doi: 10.3945/jn.114.195065. Epub 2014 Dec 3. PMID 25527677
- [Derived] Gower BA, Pollock NK, Casazza K, Clemens TL, Goree LL, Granger WM. Associations of total and undercarboxylated osteocalcin with peripheral and hepatic insulin sensitivity and beta-cell function in overweight adults. J Clin Endocrinol Metab. 2013 Jul;98(7):E1173-80. doi: 10.1210/jc.2013-1203. Epub 2013 Apr 24. PMID 23616149
- [Derived] Ellis AC, Casazza K, Chandler-Laney P, Gower BA. Higher postprandial serum ghrelin among African-American girls before puberty. J Pediatr Endocrinol Metab. 2012;25(7-8):691-6. doi: 10.1515/jpem-2012-0081. PMID 23155695
- [Derived] Ellis AC, Chandler-Laney P, Casazza K, Goree LL, Gower BA. Effects of habitual diet on ethnic differences in serum total ghrelin. Endocrine. 2012 Oct;42(2):359-65. doi: 10.1007/s12020-012-9667-2. Epub 2012 Apr 7. PMID 22481313
- [Derived] Goree LL, Chandler-Laney P, Ellis AC, Casazza K, Granger WM, Gower BA. Dietary macronutrient composition affects beta cell responsiveness but not insulin sensitivity. Am J Clin Nutr. 2011 Jul;94(1):120-7. doi: 10.3945/ajcn.110.002162. Epub 2011 May 18. PMID 21593507